CLINICAL TRIAL: NCT04374253
Title: An Open-Label, Multicenter, Rollover Study to Evaluate the Safety, Tolerability, and Efficacy of Long-Term Gantenerumab Administration in Participants With Alzheimer's Disease
Brief Title: A Study to Evaluate the Safety, Tolerability, and Efficacy of Long-Term Gantenerumab Administration in Participants With Alzheimer's Disease (AD)
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Decision to terminate development of Gantenerumab for treatment of prodromal/mild/early-stage Alzheimer's disease following results of a pre-planned analysis of the safety and efficacy of Gant in Graduate I&II (WN29922/WN39658).
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: WN42171; 2020-000766-42 (EudraCT Number)
Record Dates: First submitted 2020-05-01; First posted 2020-05-05 (Actual); Results first posted 2024-05-08 (Actual); Last update posted 2024-05-08 (Actual); Status verified 2024-04

CONDITIONS: Alzheimer Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — gantenerumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 (Experimental): Participants, who completed the double-blind part and did not enter the OLE part of Study WN29922 or WN39658, will be enrolled and receive open-label gantenerumab approximately 2 weeks after the Week 116 visit of Study WN29922 or WN39658. This will be considered the OLE baseline visit (OLE Day 1).
  Interventions: Drug: Gantenerumab
- Group 2 (Experimental): Participants, who completed the double-blind part and the OLE part of Study WN29922 or WN39658, will be enrolled and receive open-label gantenerumab approximately 2 weeks after the OLE Week 34 visit or the final dose visit in the Study WN29922 or WN39658 OLE.
  Interventions: Drug: Gantenerumab

INTERVENTIONS:
Drug: Gantenerumab — Group 1 participants who were in the active arm in the double blind part in the parent study (WN29922 or WN39658), will continue to receive open-label gantenerumab 510 mg SC, Q2W. Participants who are naive to gantenerumab treatment will be required to undergo the 3 step uptitration scheme before receiving target dose of open label gantenerumab, 510 mg SC, Q2W.
  Arms: Group 1
Drug: Gantenerumab — Group 2 participants who have completed OLE part in the parent study (WN29922 or WN39658), will continue to receive open-label gantenerumab 510 mg SC, Q2W
  Arms: Group 2

SUMMARY:
This is an open-label, multicenter, rollover study to evaluate the safety, tolerability, and efficacy of long-term administration of open-label gantenerumab in participants with AD who completed Study WN29922 or WN39658, either the double-blind or open-label extension (OLE) part.

DETAILED DESCRIPTION:
Participants who were in the active arm in the double blind part and those who have completed OLE part in the parent study, will continue receive open-label gantenerumab 510 mg sub-cutaneously (SC) every 2 weeks (Q2W). Participants who are naive to gantenerumab treatment will be required to undergo the 3 step uptitration scheme as in the parent study before receiving target dose of open label gantenerumab.

ELIGIBILITY:
Inclusion Criteria:

* Completed Study WN29922 or WN39658, either its double-blind part or OLE part, and did not discontinue study drug early
* The participant should be capable of completing assessments either alone or with the help of the caregiver
* Availability of a person (referred to as the "caregiver")
* For women of childbearing potential: agreement to remain abstinent (refrain from heterosexual intercourse) or use contraception methods with a failure rate of <1% per year (bilateral tubal ligation, male sterilization, hormonal contraceptives that inhibit ovulation, hormone-releasing intrauterine devices, and copper intrauterine devices) during the treatment period and for at least 16 weeks after the final dose of gantenerumab
* Agreement not to donate blood or blood products for transfusion for the duration of the study and for 1 year after final dose of study drug

Exclusion Criteria:

* Pregnant or breastfeeding, or intending to become pregnant during the study or within at least 16 weeks after the final dose of study drug
* Prematurely discontinued from Study WN29922 or WN39658
* Any medical condition that may jeopardize the participant's safety if he or she continues to receive study treatment
* Received any investigational treatment other than gantenerumab during or since completion of Study WN29922 or WN39658, either its double-blind or OLE part
* Evidence of disseminated leptomeningeal hemosiderosis
* Evidence of intracerebral macrohemorrhage
* Use of prohibited medication
* Evidence of ARIA-E on the last MRI scan report in Study WN29922 or WN39658, either its double-blind or OLE part

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 1382 (Actual)
Dates: Start 2021-01-26 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (268):
- United States (67):
  - Banner Alzheimer?s Institute, Phoenix, Arizona
  - Barrow Neurological Institute, Phoenix, Arizona
  - Banner Sun Health Research Insitute, Sun City, Arizona
  - Health Initiatives Research, PLLC, Fayetteville, Arkansas
  - Fullerton Neurology and Headache Center, Fullerton, California
  - Neurology Center of North Orange County, Fullerton, California
  - Irvine Center for Clinical Research, Irvine, California
  - Desert Valley Research, Redlands, California
  - Sutter Medical Group, Neurology, Sacramento, California
  - Syrentis Clinical Research, Santa Ana, California
  - California Neuroscience Research Medical Group, Inc, Sherman Oaks, California
  - Southern California Research LLC, Simi Valley, California
  - Yale University School Of Medicine, New Haven, Connecticut
  - Research Center for Clinical Studies, Inc., Norwalk, Connecticut
  - Georgetown University Medical Center, Washington D.C., District of Columbia
  - JEM Research LLC, Atlantis, Florida
  - Accel Research Sites - CRU Tampa, Bradenton, Florida
  - Bradenton Research Center, Bradenton, Florida
  - Brain Matters Research, Inc., Delray Beach, Florida
  - ClinCloud, LLC, Maitland, Florida
  - Optimus U Corp, Miami, Florida
  - Allied Biomedical Research Institute, Inc, Miami, Florida
  - Renstar Medical Research, Ocala, Florida
  - Intercoastal Medical Group, Sarasota, Florida
  - Infinity Clinical Research, LLC, Sunrise, Florida
  - Axiom Clinical Research of Florida, Tampa, Florida
  - Alzheimer?s Research and Treatment Center, Wellington, Florida
  - Emory University, Atlanta, Georgia
  - Center for Advanced Research & Education, Gainesville, Georgia
  - Southern Illinois University, School of Medicine, Springfield, Illinois
  - American Health Network Institute, LLC, Avon, Indiana
  - Fort Wayne Neurological Center, Fort Wayne, Indiana
  - Via Christi Research, Wichita, Kansas
  - Brigham and Womens Hospital; Center for Alzheimer Research & Treatment, Boston, Massachusetts
  - Boston Center for Memory, Newton, Massachusetts
  - Precise Research Centers, Flowood, Mississippi
  - University of Mississippi Medical Center, Jackson, Mississippi
  - Missouri Memory Center, Bolivar, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - University of Nebraska Medical Center; Dept of Neurological Sciences, Omaha, Nebraska
  - Cleveland Clinic Lou Ruvo; Center for Brain Research, Las Vegas, Nevada
  - The Cognitive and Research Center of New Jersey, Springfield, New Jersey
  - Advanced Memory Research Institute of NJ, Toms River, New Jersey
  - Neurological Associates of Long Island, PC, Lake Success, New York
  - Columbia University Medical Center, New York, New York
  - AD-CARE, University of Rochester Medical Center, Rochester, New York
  - Richmond Behavioral Associates, Staten Island, New York
  - SUNY Upstate Medical University, Syracuse, New York
  - Behavioral Health Research, Charlotte, North Carolina
  - Alzheimer's Memory Center, Matthews, North Carolina
  - Raleigh Neurology Associates, Raleigh, North Carolina
  - Wake Forest University, Winston-Salem, North Carolina
  - Cleveland Clinic; Cleveland Lou Ruvo Center for Brain Health ? Neurological Institute, Cleveland, Ohio
  - Ohio State University; College of Medicine, Columbus, Ohio
  - Summit Research Network Inc., Portland, Oregon
  - Abington Neurological Associates, Abington, Pennsylvania
  - The Clinical Trial Center, LLC, Jenkintown, Pennsylvania
  - Senior Adults Specialty Research, Austin, Texas
  - Kerwin Medical Center, Dallas, Texas
  - Neurology Consultants of Dallas; Research Department, Dallas, Texas
  - Alzheimers Disease & Memory Disorders Center; Department of Neurology Baylor College of Medicine, Houston, Texas
  - The University of Texas Health Science Center at Houston, Houston, Texas
  - Wasatch Clinical Research, LLC, Salt Lake City, Utah
  - University of Virginia, Charlottesville, Virginia
  - Sentara Neurology Specialists, Norfolk, Virginia
  - National Clinical Research Inc.-Richmond, Richmond, Virginia
  - UW Wisconsin-Madison, Madison, Wisconsin
- Argentina (7):
  - Hospital Italiano, CABA
  - Universidad Maimonides, Caba
  - Instituto Geriatrico Nuestra Señora de las Nieves, Capital Federal
  - Instituto Kremer, Córdoba
  - CEN Centro Especializado en Neurociencias, Córdoba
  - Instituto de Neurociencias San Agustín S.A., La Plata
  - Fundación Scherbovsky; General Department, Mendoza
- Australia (6):
  - St Vincent's Hospital Sydney; Neurology, Darlinghurst, New South Wales
  - Central Coast Neurosciences Research, Erina, New South Wales
  - Southern Neurology, Kogarah, New South Wales
  - The Queen Elizabeth Hospital; Neurology, Woodville, South Australia
  - Heidelberg Repatriation Hospital; Medical and Cognitive Research Centre, Heidelberg West, Victoria
  - Australian Alzheimer's Research Foundation, Nedlands, Western Australia
- Belgium (3):
  - AZ Sint Blasius (Dendermonde), Dendermonde
  - UZ Gent, Ghent
  - Jessa Zkh (Campus Virga Jesse), Hasselt
- Brazil (5):
  - Hospital Nossa Senhora das Graças; Setor de Pesquisa em Neurologia, Curitiba, Paraná
  - Instituto de Neurologia de Curitiba, Curitiba, Paraná
  - Clinica Clinilive ltda, Maringá, Paraná
  - Hospital das Clinicas - UFRGS, Porto Alegre, Rio Grande do Sul
  - Hospital das Clinicas - FMUSP_X; Neurologia, São Paulo, São Paulo
- Canada (7):
  - The Medical Arts Health Research Group - West Vancouver, Vancouver, British Columbia
  - Parkwood Hospital; Geriatric Medicine, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - Baycrest Health Sciences, Toronto, Ontario
  - Devonshire Clinical Research, Woodstock, Ontario
  - Center for Diagnosis and Research on Alzheimer's disease, Greenfield Park, Quebec
  - Alpha Recherche Clinique, Québec
- Chile (3):
  - Psicomed Estudios Médicos, Antofagasta
  - Biomedica Research Group, Santiago
  - Especialidades Medicas LYS, Santiago
- Beijing Tian Tan Hospital,Capital Medical University, Beijing, China
- Denmark (3):
  - Aarhus Universitetshospital; Neurologisk Afd. F, Demensklinikken, Aarhus N
  - Rigshospitalet, Hukommelsesklinikken, København Ø
  - Svendborg Sygehus; Neurologisk afdeling N, Demensklinik Fyn, Svendborg
- Finland (2):
  - Terveystalo Ruoholahti, Helsinki
  - Itä-Suomen yliopisto, Kuopion kampus, Kuopio
- France (9):
  - CHU Amiens Hopital Sud; Neurologie, Amiens Cedex1
  - Hôpital Avicenne; Centre de Recherche Clinique, Bobigny
  - Groupement Hospitalier Est - Hôpital Neurologique; Neurologie A (U502), Bron
  - CHU de la Timone - Hopital d Adultes; Service de Neurologie, Marseille
  - Hôpital Lariboisière, Paris
  - CHU Poitiers - Hopital La Miletrie, Poitiers
  - CHU Strasbourg Hôpital Hautepierre, Strasbourg
  - Gerontopole; Centre de Recherche clinique, Toulouse
  - Hopital des Charpennes, Villeurbanne
- Germany (11):
  - Ambulates Gesundheitszentrum der Charité GmbH; MVZ Neurologie Campus Benjamin Franklin, Berlin
  - ECRC Experimental and Clinical Research Center, Charité Campus Berlin Buch, Memory Clinic, Berlin
  - Universitätsklinikum Köln; Klinik und Poliklinik für Psychiatrie und Psychotherapie, Cologne
  - PANAKEIA - Arzneimittelforschung Leipzig GmbH, Leipzig
  - Universitätsmedizin derJohannes Gutenberg-Universität Mainz;Klinik für Psychiatrie und Psychotherapi, Mainz
  - Klinikum rechts der Isar der TU München; Klinik für Psychiatrie und Psychotherapie, München
  - Universitätsklinikum Münster; Klinik und Poliklinik für Neurologie, Münster
  - Universitätsklinikum Rostock Zentrum für Nervenheilkunde, Rostock
  - Universitätsklinikum Ulm; Klinik für Neurologie, Ulm
  - Studienzentrum Nordwest Dr med Joachim Springub Herr Wolfgang Schwarz, Westerstede
  - Forschungszentrum Ruhr, Witten
- Semmelweis University; Department of Neurology, Budapest, Hungary
- Italy (10):
  - Nuovo Ospedale Civile S. Agostino-Estense; Clinica Neurologica ? Dipartimento di Neuroscienze, Modena, Emilia-Romagna
  - Fondazione Santa Lucia IRCCS; Neurologia e Riabilitazione Neurologica, Rome, Lazio
  - Umberto I Policlinico di Roma-Università di Roma La Sapienza, Rome, Lazio
  - Ospedale San Giovanni Calibita Fatebenefratell;Neurologia, Rome, Lazio
  - IRCCS ?Centro S. Giovanni di Dio? Fatebenefratelli -UO Alzheimer, Brescia, Lombardy
  - IRCCS Ospedale San Raffaele; Centro Disturbi della Memoria, Milan, Lombardy
  - ASST DI MONZA; Neurologia, Monza, Lombardy
  - IRCCS Neuromed; Neurologia I-Centro studio e cura delle demenze e UVA, Pozzilli, Molise
  - AO Città della Salute e della Scienza Osp.S.Giov.Battista Molinette; SC Geriatria, Turin, Piedmont
  - Dipartimento delle Patologie Emergenti; Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo, Sicily
- Japan (34):
  - Yachiyo Hospital, Aichi
  - Nagoya Ekisaikai Hospital, Aichi
  - National Center for Geriatrics and Gerontology, Aichi
  - Medical Corporation Hakuyokai Kashiwado Hospital, Chiba
  - Tokyo Bay Advanced Medical and Makuhari Clinic, Chiba
  - Inage Neurology and Memory Clinic, Chiba
  - Juntendo University Urayasu Hospital, Chiba
  - Fukuoka University Hospital, Fukuoka
  - Southern Tohoku Medical Clinic, Fukushima
  - National Hospital Organization Hiroshima-Nishi Medical Center, Hiroshima
  - Kobe University Hospital, Hyōgo
  - Hyogo Prefectural HarimaHimeji General Medical Center, Hyōgo
  - Tsukazaki Hospital, Hyōgo
  - Matsui Dietary and Dementia Clinic, Hyōgo
  - Kagawa Prefectural Central Hospital, Kagawa
  - Shonan Kamakura General Hospital, Kanagawa
  - Rakuwakai Otowa Hospital, Kyoto
  - Uji Takeda Hospital, Kyoto
  - Okayama Kyokuto Hospital, Okayama
  - Rijikai Medical Corporation Katayama Medical Clinic, Okayama
  - MI Clinic, Osaka
  - Kishiwada Tokushukai Hospital, Osaka
  - National Hospital Organization Hizen Psychiatric Medical Center, Saga
  - NHO Shizuoka Institute of Epilepsy and Neurological Disorders, Shizuoka
  - Shizuoka City Shimizu Hospital, Shizuoka
  - Jichiidai Station Brain Clinic, Tochigi
  - Medical corporation Ichiekai Itsuki Hospital, Tokushima
  - Tokushima Hospital, Tokushima
  - Tokyo Medical and Dental University Hospital, Tokyo
  - Tokyo Medical University Hospital, Tokyo
  - Nozomi Memory Clinic, Tokyo
  - National Center of Neurology and Psychiatry, Tokyo
  - P-One Clinic, Tokyo
  - Yamagata Tokusyukai Hospital, Yamagata
- Vilnius University Hospital Santariskiu Clinics; Neurology, Vilnius, Lithuania
- Mexico (4):
  - Mexico Centre for Clinical Research, Mexico City, Mexico CITY (federal District)
  - Hospital Universitario Dr Jose Eleuterio Gonzalez UANL; Depto.de NeurologíaPta.BajaConsulta, Monterrey, Nuevo León
  - AVIX Investigación Clínica S.C, Monterrey, Nuevo León
  - Hospital Angeles de Culiacán, Neurociencias Estudios Clínicos SC, Culiacán, Sinaloa
- Brain Research Center B.V, Amsterdam, Netherlands
- Peru (3):
  - Hospital IV Alberto Sabogal Sologuren; Unidad de Investigacion, Bellavista
  - Clinica Internacional; Unidad De Investigacion, Lima
  - Hospital Nacional Dos de Mayo; Unidad de Investigacion de Neurologia, Lima
- Poland (10):
  - O?rodek Badawczo-Naukowo-Dydaktyczny Chorób Ot?piennych w ?cinawie, ?cinawa
  - Podlaskie Centrum Psychogeriatrii, Bia?ystok
  - NZOZ Vitamed, Bydgoszcz
  - NEURO-CARE Sp. z o.o. Sp. Komandytowa, Katowice
  - KO-MED Centra Kliniczne Lublin II, Lublin
  - Neurologiczny NZOZ Centrum Leczenia SM; Osrodek Badan Klinicznych, Plewiska
  - Senior Sp. Z O.O. Poradnia Psychogeriatryczna, Sopot
  - mMED Maciej Czarnecki, Warsaw
  - Pratia S.A., Warsaw
  - NZOZ WCA, Wroc?aw
- Portugal (4):
  - Hospital de Braga; Servico de Neurologia, Braga
  - HUC; Servico de Neurologia, Coimbra
  - Hospital da Senhora da Oliveira-Guimarães; Serviço de Neurologia, Guimarães
  - Hospital Geral de Santo Antonio; Servico de Neurologia, Porto
- Puerto Rico (2):
  - Santa Cruz Behavioral PSC, Bayamón
  - University of Puerto Rico - Medical Science Campus; Internal Medicine, San Juan
- Russia (9):
  - FSBHI Siberian Clinical Center of the Federal Medical and Biological Agency, Krasnoyarsk, Krasnoyarsk Krai
  - University ?linic of headaches, Moscow, Moscow Oblast
  - City Clin Hosp n.a. S.P.Botkin, Moscow, Moscow Oblast
  - City Polyclinic No. 2 of the Department of Healthcare of the City of Moscow, Moskva, Moscow Oblast
  - FSBMEI HPE "Military Medical Academy n.a. S.M. Kirov" of the MoD of the RF, Saint Petersburg, Sankt-Peterburg
  - Vertebronevrologiya LLC, Kazan', Tatarstan Republic
  - State autonomous institution of healthcare Inter-regional clinical and diagnostic center, Kazan', Tatarstan Republic
  - MHI City Clinical Hospital #2 named after V.I. Razumovsky; Psychiatric, Saratov
  - Nebbiolo Center for Clinical Trials, Tomsk
- South Korea (11):
  - Dong-A University Hospital, Busan
  - Myongji Hospital, Gyeonggi-do
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Seoul National University Bundang Hospital, Seongnam-si
  - Hanyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul St Mary's Hospital, Seoul
  - Ewha Womans University Hospital (Seoul), Seoul
- Spain (32):
  - Hospital General Universitario de Elche; Servicio de Neurología, Elche, Alicante
  - Hospital Universitari de Bellvitge; Servicio de Neurologia, L'Hospitalet de Llobregat, Barcelona
  - Hospital General De Catalunya; Servicio de Neurologia, Sant Cugat del Vallès, Barcelona
  - Hospital Mutua De Terrasa; Servicio de Neurologia, Terrassa, Barcelona
  - Hospital Virgen del Puerto. Servicio de Neurología, Plasencia, Caceres
  - Hospital Universitario Marques de Valdecilla; Servicio de Neurología, Santander, Cantabria
  - Policlínica Guipuzcoa; Servicio de Neurología, Donostia / San Sebastian, Guipuzcoa
  - Hospital San Pedro; Servicio de Neurología, Logroño, La Rioja
  - Hospital Universitario de Santa Maria; Servicio de Neurología, Lleida, Lerida
  - HM Universitario Puerta del Sur CINAC (C.Integ.Neuroc);; Servicio de Psiquiatría, Móstoles, Madrid
  - Hospital Quiron de Madrid; Servicio de Neurologia, Pozuelo de Alarcón, Madrid
  - Clinica Universitaria de Navarra; Servicio de Neurología, Pamplona, Navarre
  - Clinica Universitaria de Navarra, Pamplona, Navarre
  - CAE OROITU; Servicio de Neurología, Getxo, Vizcaya
  - Hospital General Universitario de Albacete; Servicio de Neurología, Albacete
  - Hospital del Mar; Servicio de Neurologia, Barcelona
  - Fundación ACE; Servicio de Neurología, Barcelona
  - Hospital Vall d'Hebron; Servicio de Neurología, Barcelona
  - Hospital Clinic i Provincial; Servicio de Neurologia, Barcelona
  - Hospital de la Santa Creu i Sant Pau; Servicio de Neurologia, Barcelona
  - Hospital Universitario Reina Sofia; Servicio de Neurologia, Córdoba
  - Universitario de La Princesa; Servicio de Neurología, Madrid
  - Hospital Ramon y Cajal; Servicio de Neurologia, Madrid
  - Hospital Ruber Internacional; Servicio de Neurología, Madrid
  - Hospital Universitario 12 de Octubre; Servicio de Neurologia, Madrid
  - Complejo Asistencial Universitario de Salamanca; Servicio de Psiquiatría, Salamanca
  - Hospital Virgen del Rocío; Servicio de Neurología, Seville
  - Hospital Victoria Eugenia; Servico Neurología, Seville
  - Hospital Universitario Dr. Peset; Servicio de Neurologia, Valencia
  - Hospital Universitario la Fe; Servicio de Neurologia, Valencia
  - Complejo Asistencial de Zamora; Servicio Psiquiatria, Zamora
  - Servicio de Neurología Hospital Viamed Montecanal., Zaragoza
- Sweden (3):
  - Skånes Universitetssjukhus Malmö, Minneskliniken, Malmo
  - Sahlgrenska Academy University,Neuroscience and Physiology;Departmt of Psychiatry and Neurochemistry, Mölndal
  - KAROLINSKA UNI HOSPITAL, HUDDINGE; Mottagning Kognitiv Forskning, M54, Stockholm
- Taiwan (6):
  - Changhua Christian Hospital; Neurology, Changhua County
  - Kaohsiung Medical University Hospital; Neurology, Kaohsiung City
  - Chang Gung Memorial Foundation - Kaohsiung - Neurology, Niaosong Dist.
  - China Medical University Hospital; Neurology, North Dist.
  - National Taiwan University Hospital; Neurology, Taipei
  - Chang Gung Memorial Foundation - Linkou - Neurology, Taoyuan District
- Ondokuz Mayis Univ. Med. Fac.; Neurology, Samsun, Turkey (Türkiye)
- United Kingdom (12):
  - The Rice Centre; Royal United Hospital, Bath
  - Re:Cognition Health Birmingham, Birmingham
  - The Fritchie Centre, Charlton Lane Centre, Charlon Lane, Leckhampton; The Fritchie Centre, Cheltenham
  - Surrey and Borders NHS Foundation Trust; Research and Development Department, Chertsey
  - Ninewells Hospital, Dundee
  - Queen Elizabeth University Hospital - PPDS, Glasgow
  - St George?s Hospital, London
  - Re:Cognition Health London, London
  - Charing Cross Hospital, London
  - Campus for Ageing and Vitality, Newcastle
  - Royal Hallamshire Hospital Sheffield Teaching Hospitals NHS Foundation Trust, Sheffield
  - University Southampton NHS Foundation Trust; Wessex Neurologica Centre, Southampton

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Salloway S, Wojtowicz J, Voyle N, Lane CA, Klein G, Lyons M, Rossomanno S, Mazzo F, Bullain S, Barkhof F, Bittner T, Schneider A, Grundman M, Aldea R, Boada M, Smith J, Doody R. Amyloid-Related Imaging Abnormalities (ARIA) in Clinical Trials of Gantenerumab in Early Alzheimer Disease. JAMA Neurol. 2025 Jan 1;82(1):19-29. doi: 10.1001/jamaneurol.2024.3937. PMID 39556389

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in this study at 258 investigative centers across 28 countries from 26 January 2021 to 06 March 2023. A total of 1382 participants who completed either the double-blind (DB) part or open-label extension (OLE) part in parent GRADUATE studies WN29922 (NCT03444870) or WN39658 (NCT03443973) were enrolled in this study to receive open-label gantenerumab.
Pre-assignment Details: Participants who completed DB and OLE part received gantenerumab approximately 2 weeks after OLE Week 34 visit or final OLE dose visit in the parent study. Participants who completed DB part and did not enter the OLE part received gantenerumab approximately 2 weeks after the Week 116 visit of the parent study.
Groups:
- Placebo: Participated in Graduate OLE: Participants treated with placebo in the DB part and who completed the DB and OLE up titration in study WN29922 (GRADUATE I) or WN39658 (GRADUATE II), continued receiving open-label gantenerumab, 510 milligrams (mg), SC, every two weeks (Q2W).
- Placebo: No Participation in Graduate OLE: Participants treated with placebo in the DB part and who did not enter the OLE part of study WN29922 (GRADUATE I) or WN39658 (GRADUATE II) received gantenerumab SC injections with gradual up titration starting at a dose of 120 mg, every four weeks (Q4W) for 3 doses, followed by 255 mg, Q4W for 3 doses, and then at a dose of 510 mg, Q4W for 3 doses before receiving open-label gantenerumab, 510 mg SC injections, Q2W. To maintain the blind to previous treatment assignment, participants received Q2W, SC injections, with alternate doses containing gantenerumab matching placebo.
- Gantenerumab: Participated in Graduate OLE: Participants treated with gantenerumab in the DB part and who completed the DB and OLE part of study WN29922 (GRADUATE I) or WN39658 (GRADUATE II) continued receiving open-label gantenerumab, 510 mg, SC, Q2W.
- Gantenerumab: No Participation in Graduate OLE: Participants treated with gantenerumab in the DB part and who did not enter the OLE part of study WN29922 (GRADUATE I) or WN39658 (GRADUATE II) continued receiving open-label gantenerumab 510 mg SC, Q2W.
Period: Overall Study
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Started | 15 | 696 | 28 | 643
Safety-evaluable (SE) Analysis Set (SE analysis set included all participants enrolled who received at least one dose of study drug in this study or in the OLE part of the parent studies (GRADUATE I or GRADUATE II). Six participants randomized to placebo arm during the double-blind treatment in the parent studies received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety evaluable set.) | 14 | 691 | 29 | 647
Intent-to-Treat Analysis (ITT) Set (ITT analysis set included all enrolled participants who received at least one dose of study drug. Participants will be analyzed by the treatment they were randomized to in the parent studies (GRADUATE I or GRADUATE II).) | 15 | 696 | 28 | 642
Magnetic Resonance Imaging (MRI) SE (M-SE) Analysis Set (M-SE analysis set included all participants in the SE analysis set who had at least one post-baseline safety MRI scan.) | 14 | 671 | 29 | 627
Completed | 0 | 0 | 0 | 0
Not Completed | 15 | 696 | 28 | 643
Not completed — Adverse Event | 0 | 26 | 2 | 12
Not completed — Study terminated by sponsor | 13 | 593 | 21 | 567
Not completed — Withdrawal by Subject | 0 | 55 | 3 | 40
Not completed — Physician Decision | 1 | 10 | 1 | 10
Not completed — Protocol Violation | 0 | 0 | 0 | 2
Not completed — Death | 0 | 3 | 1 | 1
Not completed — Lack of Efficacy | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 1 | 1 | 0 | 2
Not completed — Reason Not Specified | 0 | 8 | 0 | 8

BASELINE CHARACTERISTICS:
Population: ITT analysis set included all enrolled participants, who received at least one dose of study drug. Participants were analyzed by the treatment they were randomized to in the parent studies (GRADUATE I or GRADUATE II).
Groups:
- Placebo: Participated in Graduate OLE: Participants treated with placebo in the DB part and who completed the DB and OLE up titration in study WN29922 (GRADUATE I) or WN39658 (GRADUATE II), continued receiving open-label gantenerumab, 510 mg, SC, Q2W.
- Placebo: No Participation in Graduate OLE: Participants treated with placebo in the DB part and who did not enter the OLE part of study WN29922 (GRADUATE I) or WN39658 (GRADUATE II) received gantenerumab SC injections with gradual up titration starting at a dose of 120 mg, Q4W for 3 doses, followed by 255 mg, Q4W for 3 doses, and then at a dose of 510 mg, Q4W for 3 doses before receiving open-label gantenerumab, 510 mg SC injections, Q2W. To maintain the blind to previous treatment assignment, participants received Q2W, SC injections, with alternate doses containing gantenerumab matching placebo.
- Total: Total of all reporting groups
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE | Total
Number analyzed (Participants) | 15 | 696 | 28 | 642 | 1381
Age, Continuous [Mean (Standard Deviation); unit: years] | 76.7 (7.8) | 73.6 (7.4) | 74.1 (8.0) | 73.0 (7.7) | 73.4 (7.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 387 | 14 | 382 | 794
  Male | 4 | 309 | 14 | 260 | 587
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 6 | 116 | 14 | 89 | 225
  Not Hispanic or Latino | 9 | 576 | 14 | 548 | 1147
  Unknown or Not Reported | 0 | 4 | 0 | 5 | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 25 | 4 | 18 | 47
  Asian | 1 | 104 | 1 | 87 | 193
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 6 | 0 | 4 | 10
  White | 14 | 549 | 22 | 518 | 1103
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 12 | 1 | 15 | 28

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least One Adverse Event (AE) and Serious Adverse Event (SAE)
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of casual attribution. A SAE is any AE that is fatal, life threatening, requires or prolongs inpatient hospitalization, results in persistent or significant disability/incapacity, is a congenital anomaly/birth defect in a neonate/infant born to a mother exposed to study drug or a significant medical event in the investigator's judgment. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: From Baseline (OLE Day 1) up to 14 weeks after the last dose (up to 134 weeks)
Population: SE analysis set included all participants enrolled who received at least one dose of study drug in this study or in the OLE part of the parent studies (GRADUATE I or GRADUATE II). Six participants randomized to placebo arm during the double-blind treatment in the parent studies received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety evaluable set.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 14 | 691 | 29 | 647
Participants
  AEs | 13 | 510 | 25 | 487
  SAEs | 2 | 72 | 4 | 54

2. Primary Outcome: Number of Participants With Post-baseline Suicidal Ideation or Suicidal Behavior as Measured Using Columbia-Suicide Severity Rating Scale (C-SSRS) Score
Description: C-SSRS= assesses lifetime suicidality of participant (at baseline) & any new instances of suicidality (since last visit). Structured interview prompts recollection of suicidal ideation (intensity of ideation, behavior, & attempts with actual/potential lethality). Categories have yes/no responses, include Wish to be Dead; Non-specific Active Suicidal Thoughts; Active Suicidal Ideation with Any Methods (Not Plan) without Intent to Act; Active Suicidal Ideation with Some Intent to Act, without Specific Plan; Active Suicidal Ideation with Specific Plan and Intent, Preparatory Acts and Behavior; Aborted/Interrupted Attempt; Actual Attempt (non-fatal); Completed Suicide. Suicidal ideation/behavior= "yes" to any of listed categories. Score of 0= no suicide risk. Score of 1 or higher= suicidal ideation or behavior. Categories with non-zero values are only reported here. First dosing visit in OLE (first dosing in current study or OLE period of parent GRADUATE studies)=baseline (OLE Day 1).
Time Frame: From Baseline (OLE Day 1) up to 14 weeks after the last dose (up to 134 weeks)
Population: SE analysis set included all participants enrolled who received at least one dose of study drug in this study or in the OLE part of the parent studies. Six participants randomized to placebo arm during the double-blind treatment in the parent studies received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety evaluable set. Overall number analyzed is the number of participants with data available for analyses.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 14 | 631 | 29 | 588
Participants
  Suicidal Ideation: Passive | 1 | 11 | 1 | 11
  Suicidal Ideation: Active-Nonspecific (No Method, Intent, or Plan) | 0 | 3 | 0 | 2
  Suicidal Ideation: Active-Method, but No Intent or Plan | 1 | 0 | 1 | 0
  Suicidal Ideation: No event | 12 | 617 | 27 | 575
  Suicidal Behavior: Completed Suicide | 0 | 0 | 0 | 2
  Suicidal Behavior: Aborted Attempt | 0 | 1 | 0 | 0
  Suicidal Behavior: Preparatory Actions Toward Imminent Suicidal Behaviors | 0 | 1 | 0 | 0
  Suicidal Behavior: No event | 14 | 629 | 29 | 586
  Self-injurious Behavior, Without Suicidal Intent: Self-Injurious Behavior - No Suicidal Intent | 0 | 2 | 0 | 0
  Self-Injurious Behavior Without Suicidal Intent: No event | 14 | 629 | 29 | 588

3. Primary Outcome: Number of Participants With at Least One Amyloid-Related Imaging Abnormalities-Edema (ARIA-E) Confirmed by MRI
Description: ARIA are an identified risk with anti-amyloid antibodies, including gantenerumab. These changes can be identified on brain MRI. In ARIA-E, (E for oedema or effusion), oedema can be seen in different areas of the brain on MRI, representing fluid leakage into the brain parenchyma or sulcal spaces. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: From Baseline (OLE Day 1) up to 14 weeks after the last dose (up to 134 weeks)
Population: M-SE analysis set included all participants in the SE analysis set who had at least one post-baseline safety MRI scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 14 | 671 | 29 | 627
Participants | 6 | 104 | 5 | 27

4. Primary Outcome: Number of Participants With at Least One Amyloid-Related Imaging Abnormalities-Haemosiderin Deposition (ARIA-H) Confirmed by MRI
Description: ARIA are an identified risk with anti-amyloid antibodies, including gantenerumab. These changes can be identified on brain MRI. ARIA-H (H for hemosiderosis) are small foci of signal loss observed on MRI sequences sensitive for paramagnetic tissue properties and comprise cerebral microbleeds (small foci of bleeding in the brain parenchyma) and leptomeningeal hemosiderosis (small foci of bleeding on the surface of the brain). These changes also occur sporadically in AD. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: From Baseline (OLE Day 1) up to 14 weeks after the last dose (up to 134 weeks)
Population: M-SE analysis set included participants in the SE analysis set who had at least one post-baseline safety MRI scan.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 14 | 671 | 29 | 627
Participants | 3 | 85 | 4 | 40

5. Primary Outcome: Number of Participants With Injection-Site Reactions (ISRs)
Description: An AE is any unfavorable and unintended sign, symptom, or disease temporally associated with the use of a pharmaceutical product, regardless of casual attribution. Local injection reactions (or injection site reactions) are defined as AEs related to the injection site that occur during or within 24 hours after study drug administration that are judged to be related to the study drug injection. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: From Baseline (OLE Day 1) up to 14 weeks after the last dose (up to 134 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 14 | 691 | 29 | 647
Participants | 3 | 63 | 1 | 80

6. Primary Outcome: Number of Participants Who Discontinued the Study Due an AE
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of casual attribution. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: From Baseline (OLE Day 1) up to 14 weeks after the last dose (up to 134 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 14 | 691 | 29 | 647
Participants | 0 | 9 | 1 | 7

7. Primary Outcome: Number of Participants With at Least One Adverse Event of Special Interest (AESI)
Description: An AE is any untoward medical occurrence in a clinical investigation participant administered a pharmaceutical product, regardless of casual attribution. AEs that were considered to be of special interest for this study included cases of potential drug-induced liver injury that include an elevated ALT or AST in combination with either an elevated bilirubin or clinical jaundice, as defined by Hy's Law and suspected transmission of an infectious agent by the study drug. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: From Baseline (OLE Day 1) up to 14 weeks after the last dose (up to 134 weeks)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 14 | 691 | 29 | 647
Participants | 0 | 0 | 0 | 0

8. Secondary Outcome: Change From Baseline Over Time in Clinical Dementia Rating - Global Score (CDR-GS)
Description: CDR was derived through semi-structured interview with the participant and an appropriate informant, and it rated impairment across six domains: memory, orientation, judgment, and problem solving, community affairs, home and hobbies, and personal care on a 5-point scale for which 0=normal, 0.5=very mild dementia, 1=mild dementia, 2=moderate dementia, and 3= severe dementia. The score range for the CDR-GS is from 0 to 3 and a high score on the CDR-GS would indicate a high disease severity. A negative change from baseline indicates improvement. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: Baseline (OLE Day 1), Weeks 24, 36, 52, 76 and 104
Population: ITT analysis set included all enrolled participants, who received at least one dose of study drug. Participants will be analyzed by the treatment they were randomized to in the parent studies (GRADUATE I or GRADUATE II). Overall number analyzed is the number of participants with data available for analyses. The number of participants analyzed indicates the number of participants with data available for analyses at the specified timepoint.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 15 | 693 | 25 | 641
score on a scale
  Change from Baseline at Week 24: number analyzed (Participants) | 15 | 611 | 25 | 561
  Change from Baseline at Week 24 | 0.4 (0.50) | 0.1 (0.43) | 0.1 (0.53) | 0.1 (0.41)
  Change from Baseline at Week 36: number analyzed (Participants) | 5 | 107 | 9 | 89
  Change from Baseline at Week 36 | 0.4 (0.55) | 0.3 (0.55) | 0.1 (0.42) | 0.2 (0.47)
  Change from Baseline at Week 52: number analyzed (Participants) | 14 | 336 | 20 | 327
  Change from Baseline at Week 52 | 0.3 (0.46) | 0.2 (0.44) | -0.1 (0.43) | 0.2 (0.46)
  Change from Baseline at Week 76: number analyzed (Participants) | 11 | 169 | 19 | 161
  Change from Baseline at Week 76 | 0.5 (0.69) | 0.3 (0.47) | 0.2 (0.75) | 0.3 (0.44)
  Change from Baseline at Week 104: number analyzed (Participants) | 5 | 19 | 13 | 20
  Change from Baseline at Week 104 | 0.6 (0.89) | 0.6 (0.52) | 0.2 (0.43) | 0.3 (0.50)

9. Secondary Outcome: Change From Baseline Over Time in Clinical Dementia Rating (CDR) - Sum of Boxes (SB)
Description: CDR was derived through semi-structured interview with the participant and an appropriate informant, and it rated impairment across six domains: memory, orientation, judgment, and problem solving, community affairs, home and hobbies, and personal care on a 5-point scale for which 0=no impairment, 0.5=questionable impairment, and 1, 2, and 3=mild, moderate, and severe impairment, respectively. The CDR-SB is based on summing each of the domain box scores with total score ranging from 0-18 with higher scores reflecting greater cognitive and functional impairment. A negative change from baseline indicates improvement. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: Baseline (OLE Day 1), Weeks 24, 36, 52, 76 and 104
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 15 | 693 | 28 | 641
score on a scale
  Change from Baseline at Week 24: number analyzed (Participants) | 15 | 611 | 25 | 561
  Change from Baseline at Week 24 | 2.10 (2.473) | 0.83 (1.787) | 1.00 (2.529) | 0.70 (1.754)
  Change from Baseline at Week 36: number analyzed (Participants) | 5 | 107 | 9 | 89
  Change from Baseline at Week 36 | 2.90 (2.608) | 1.39 (2.397) | 0.72 (2.265) | 1.11 (2.161)
  Change from Baseline at Week 52: number analyzed (Participants) | 14 | 336 | 20 | 327
  Change from Baseline at Week 52 | 2.57 (2.286) | 1.60 (1.906) | 0.80 (1.351) | 1.50 (2.051)
  Change from Baseline at Week 76: number analyzed (Participants) | 11 | 169 | 19 | 161
  Change from Baseline at Week 76 | 2.68 (3.133) | 2.20 (1.994) | 1.95 (3.218) | 1.97 (2.249)
  Change from Baseline at Week 104: number analyzed (Participants) | 5 | 19 | 13 | 20
  Change from Baseline at Week 104 | 3.80 (3.213) | 3.26 (2.751) | 1.15 (2.470) | 1.80 (1.949)

10. Secondary Outcome: Change From Baseline Over Time in Mini-Mental State Examination (MMSE) Score
Description: MMSE is a rater-administered performance-based outcome (PerfO) that includes a set of standardized questions used to evaluate possible cognitive impairment and help stage the severity level of this impairment. The questions target six areas: orientation, registration, attention, short-term recall, language, and constructional praxis/visuospatial abilities. Total score ranges from 0-30, with lower scores indicating greater impairment. A positive change from baseline indicates improvement. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: Baseline (OLE Day 1), Weeks 24, 36, 52, 76 and 104
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 15 | 694 | 28 | 641
score on a scale
  Change from Baseline at Week 24: number analyzed (Participants) | 15 | 622 | 27 | 571
  Change from Baseline at Week 24 | -0.3 (2.41) | -1.2 (2.87) | -0.9 (2.39) | -1.1 (2.69)
  Change from Baseline at Week 36: number analyzed (Participants) | 5 | 111 | 9 | 93
  Change from Baseline at Week 36 | -1.8 (3.35) | -1.6 (2.83) | -0.3 (1.66) | -1.7 (3.18)
  Change from Baseline at Week 52: number analyzed (Participants) | 15 | 346 | 21 | 337
  Change from Baseline at Week 52 | -1.9 (2.94) | -2.3 (3.15) | -2.0 (3.49) | -2.1 (3.14)
  Change from Baseline at Week 76: number analyzed (Participants) | 12 | 173 | 20 | 165
  Change from Baseline at Week 76 | -2.9 (3.20) | -3.2 (3.39) | -2.9 (3.97) | -3.0 (3.56)
  Change from Baseline at Week 104: number analyzed (Participants) | 5 | 19 | 14 | 21
  Change from Baseline at Week 104 | -3.6 (5.13) | -4.3 (3.93) | -2.9 (3.92) | -3.0 (4.12)

11. Secondary Outcome: Change From Baseline Over Time in Alzheimer Disease Assessment Scale-Cognition, Subscale 11 (ADAS-Cog11) Score
Description: ADAS-Cog11 was designed to measure cognitive symptom change in participants with Alzheimer's Disease (AD) and consisted of 11 tasks. The standard 11 items (and corresponding score range) were: word recall (0-10), commands (0-5), constructional praxis (0-5), naming objects and fingers (0-5), ideational praxis (0-5), orientation (0-8), word recognition (0-12), spoken language ability (0-5), comprehension of spoken language (0-5), word-finding difficulty (0-5), and remembering test instructions (0-5). The test included 7 performance items and 4 clinician-rated items. The ADAS-Cog11 total score was the sum of all 11 individual items, with a total score ranging from 0 (no impairment) to 70 (severe impairment). Higher scores indicated more severe cognitive impairment. A negative change from baseline indicates improvement. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: Baseline (OLE Day 1), Weeks 24, 36, 52, 76 and 104
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 14 | 688 | 28 | 630
score on a scale
  Change from Baseline at Week 24: number analyzed (Participants) | 14 | 611 | 27 | 549
  Change from Baseline at Week 24 | 2.4 (5.56) | 2.4 (5.47) | 1.6 (5.29) | 2.8 (5.22)
  Change from Baseline at Week 36: number analyzed (Participants) | 5 | 107 | 9 | 86
  Change from Baseline at Week 36 | 12.0 (10.00) | 3.9 (6.80) | -3.7 (5.50) | 4.0 (5.46)
  Change from Baseline at Week 52: number analyzed (Participants) | 14 | 332 | 20 | 326
  Change from Baseline at Week 52 | 5.6 (9.55) | 3.7 (6.13) | 1.9 (5.89) | 4.7 (6.61)
  Change from Baseline at Week 76: number analyzed (Participants) | 11 | 170 | 20 | 162
  Change from Baseline at Week 76 | 6.6 (10.90) | 5.9 (7.52) | 7.0 (9.50) | 6.1 (7.80)
  Change from Baseline at Week 104: number analyzed (Participants) | 5 | 19 | 13 | 22
  Change from Baseline at Week 104 | 8.4 (14.12) | 7.8 (7.65) | 3.8 (6.67) | 8.2 (10.26)

12. Secondary Outcome: Change From Baseline Over Time in Alzheimer Disease Assessment Scale-Cognition, Subscale 13 (ADAS-Cog13) Score
Description: The ADAS-Cog13 total score includes all of the items in the ADAS-Cog11 in addition to delayed word recall and the number cancellation. For the ADAS-cog 13 the range is 0-85 (score range for Delayed Word Recall [DWR] score is 0-10 and for Number Cancellation [NC] is 0-5, thus the score is ADAS-cog 11[0-70] plus the scores for DWR and NC). A higher score indicates worse performance. A negative change from baseline indicates improvement in cognitive function. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: Baseline (OLE Day 1), Weeks 24, 36, 52, 76 and 104
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 14 | 677 | 28 | 623
score on a scale
  Change from Baseline at Week 24: number analyzed (Participants) | 14 | 597 | 27 | 542
  Change from Baseline at Week 24 | 2.9 (6.29) | 3.0 (5.73) | 2.0 (5.53) | 3.3 (5.45)
  Change from Baseline at Week 36: number analyzed (Participants) | 5 | 104 | 9 | 84
  Change from Baseline at Week 36 | 13.2 (11.52) | 4.7 (7.05) | -3.4 (5.39) | 4.7 (5.85)
  Change from Baseline at Week 52: number analyzed (Participants) | 14 | 325 | 20 | 319
  Change from Baseline at Week 52 | 6.7 (10.13) | 4.3 (6.45) | 2.7 (6.01) | 5.3 (6.94)
  Change from Baseline at Week 76: number analyzed (Participants) | 11 | 164 | 20 | 161
  Change from Baseline at Week 76 | 7.9 (11.89) | 6.8 (7.85) | 7.7 (9.76) | 6.7 (8.22)
  Change from Baseline at Week 104: number analyzed (Participants) | 5 | 19 | 13 | 22
  Change from Baseline at Week 104 | 10.4 (14.98) | 8.7 (8.13) | 4.8 (6.74) | 8.8 (10.22)

13. Secondary Outcome: Change From Baseline Over Time in Verbal Fluency Task Score
Description: VFT is a rater administered PerfO that measures speed and flexibility of verbal thought with a total score that ranges from 0-99 (lower scores indicating lower performance). A positive change from baseline indicates improvement. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: Baseline (OLE Day 1), Weeks 24, 36, 52, 76 and 104
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 15 | 693 | 28 | 641
score on a scale
  Change from Baseline at Week 24: number analyzed (Participants) | 15 | 622 | 27 | 567
  Change from Baseline at Week 24 | 0.2 (2.73) | -0.9 (3.15) | -1.0 (2.83) | -0.6 (4.73)
  Change from Baseline at Week 36: number analyzed (Participants) | 5 | 108 | 9 | 90
  Change from Baseline at Week 36 | -2.2 (3.42) | -1.2 (3.07) | -0.6 (2.70) | -1.4 (3.45)
  Change from Baseline at Week 52: number analyzed (Participants) | 15 | 346 | 20 | 337
  Change from Baseline at Week 52 | -1.5 (3.02) | -1.5 (3.60) | -0.4 (2.39) | -1.5 (5.77)
  Change from Baseline at Week 76: number analyzed (Participants) | 12 | 176 | 19 | 164
  Change from Baseline at Week 76 | -1.3 (2.83) | -2.1 (3.66) | -1.3 (4.36) | -2.8 (7.54)
  Change from Baseline at Week 104: number analyzed (Participants) | 5 | 19 | 13 | 21
  Change from Baseline at Week 104 | -0.6 (4.22) | -3.8 (3.79) | -0.8 (4.09) | -3.3 (2.50)

14. Secondary Outcome: Change From Baseline Over Time in Coding (Digit Symbol Substitution Test [DSST]) Subset
Description: Coding, also called DSST is a rater administered PerfO that measures speed of processing and associative memory with a total score that ranges from 0-135 (lower scores indicating lower performance). The DSST was adapted from the Wechsler Adult Intelligence Scale. The 120-second version of the test was used in this study. Positive change from baseline indicates improvement. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: Baseline (OLE Day 1), Weeks 24, 36, 52, 76 and 104
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 15 | 693 | 28 | 640
score on a scale
  Change from Baseline at Week 24: number analyzed (Participants) | 14 | 617 | 27 | 563
  Change from Baseline at Week 24 | -0.5 (6.31) | -2.8 (7.84) | -0.3 (9.02) | -2.3 (8.04)
  Change from Baseline at Week 36: number analyzed (Participants) | 5 | 107 | 9 | 89
  Change from Baseline at Week 36 | -8.0 (10.00) | -4.8 (8.09) | 6.2 (13.96) | -3.0 (9.66)
  Change from Baseline at Week 52: number analyzed (Participants) | 15 | 343 | 20 | 333
  Change from Baseline at Week 52 | -3.1 (7.61) | -5.0 (8.60) | -2.8 (14.00) | -4.7 (8.79)
  Change from Baseline at Week 76: number analyzed (Participants) | 11 | 171 | 19 | 164
  Change from Baseline at Week 76 | -3.4 (8.49) | -7.2 (10.12) | -7.1 (8.99) | -6.0 (9.71)
  Change from Baseline at Week 104: number analyzed (Participants) | 5 | 19 | 13 | 21
  Change from Baseline at Week 104 | 0.4 (9.94) | -4.5 (13.25) | -5.2 (11.95) | -7.0 (11.04)

15. Secondary Outcome: Change in Functional Activities Questionnaire (FAQ) Score
Description: FAQ is a rater-administered observer-reported outcome (ObsRO) (informant-based measure) that measures a participant's functional ability to perform complex higher-order activities. The observer provides performance ratings of the target person on ten complex higher-order activities. Total score that ranges from 0-30, with higher scores reflecting greater functional impairment. A negative change from baseline indicates improvement. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: Baseline (OLE Day 1), Weeks 24, 36, 52, 76 and 104
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 15 | 694 | 27 | 637
score on a scale
  Change from Baseline at Week 24: number analyzed (Participants) | 15 | 618 | 25 | 568
  Change from Baseline at Week 24 | 1.2 (4.04) | 1.6 (4.36) | 0.1 (3.15) | 1.5 (4.09)
  Change from Baseline at Week 36: number analyzed (Participants) | 5 | 111 | 9 | 96
  Change from Baseline at Week 36 | -1.0 (1.87) | 2.7 (5.07) | 1.3 (6.18) | 1.7 (4.92)
  Change from Baseline at Week 52: number analyzed (Participants) | 14 | 346 | 19 | 333
  Change from Baseline at Week 52 | 2.1 (3.80) | 2.6 (4.39) | 2.7 (3.73) | 2.6 (4.81)
  Change from Baseline at Week 76: number analyzed (Participants) | 13 | 172 | 20 | 162
  Change from Baseline at Week 76 | 2.3 (3.66) | 4.0 (4.55) | 3.3 (3.95) | 3.5 (5.12)
  Change from Baseline at Week 104: number analyzed (Participants) | 5 | 17 | 13 | 21
  Change from Baseline at Week 104 | 3.2 (4.92) | 4.5 (4.09) | 4.1 (4.91) | 1.7 (5.07)

16. Secondary Outcome: Change in Alzheimer Disease Cooperative Study Group-Activities of Daily Living (ADCS-ADL) Score
Description: ADCS-ADL is a 23-item rater-administered, ObsRO that captures a participant's ability to perform basic activities of daily living (e.g., eating and toileting) and more complex ADL or instrumental activities of daily living (iADL, e.g., using the telephone, managing finances, preparing a meal). Total score ranges from 0-78, with higher scores reflecting better functioning. A positive change from baseline indicates improvement. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: Baseline (OLE Day 1), Weeks 24, 36, 52, 76 and 104
Population: as for outcome 8
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 15 | 694 | 27 | 639
score on a scale
  Change from Baseline at Week 24: number analyzed (Participants) | 15 | 618 | 25 | 569
  Change from Baseline at Week 24 | -4.7 (5.15) | -2.9 (7.07) | -2.0 (7.10) | -3.2 (6.69)
  Change from Baseline at Week 36: number analyzed (Participants) | 4 | 111 | 9 | 96
  Change from Baseline at Week 36 | -12.5 (12.40) | -5.6 (9.55) | -2.1 (6.23) | -4.9 (8.53)
  Change from Baseline at Week 52: number analyzed (Participants) | 14 | 344 | 19 | 334
  Change from Baseline at Week 52 | -9.4 (7.49) | -5.9 (8.97) | -4.4 (8.09) | -6.2 (8.38)
  Change from Baseline at Week 76: number analyzed (Participants) | 13 | 172 | 20 | 162
  Change from Baseline at Week 76 | -10.8 (11.19) | -7.8 (9.87) | -8.3 (11.22) | -6.9 (9.62)
  Change from Baseline at Week 104: number analyzed (Participants) | 5 | 17 | 13 | 21
  Change from Baseline at Week 104 | -11.6 (17.99) | -6.6 (10.20) | -6.3 (13.52) | -9.9 (12.21)

17. Secondary Outcome: Number of Participants With Anti-drug Antibody (ADA) to Gantenerumab
Description: The number of participants with positive results for ADA against gantenerumab at any of the post-baseline assessment time-points were reported. Evaluable participant during OLE was participant with an ADA assay result from at least one sample during OLE. Treatment Emergent ADA = A participant with a negative or missing baseline ADA result(s) and at least one positive post-baseline ADA result. The first dosing visit in the OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Time Frame: From Baseline (OLE Day 1) up to 14 weeks after the last dose (up to 134 weeks)
Population: SE analysis set: all participants enrolled who received at least one dose of study drug in this study or in OLE part of parent studies (GRADUATE I or GRADUATE II). Six participants randomized to placebo arm during the double-blind treatment in the parent studies received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety evaluable set. Overall number analyzed is the number of participants with an ADA assay result from any post-baseline sample.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
Number analyzed (Participants) | 14 | 656 | 29 | 617
Participants | 1 | 17 | 1 | 14

ADVERSE EVENTS:
Time Frame: From Baseline (OLE Day 1) up to 14 weeks after the last dose (up to 134 weeks)
Description: All-cause mortality and Adverse events: SE analysis set. Six participants randomized to placebo arm during the double-blind treatment in the parent studies received at least one dose of gantenerumab and were considered in the gantenerumab arm for safety evaluable set. First dosing visit in OLE (first dosing in current study or first dosing in the OLE period of the parent GRADUATE studies) was considered as baseline (OLE Day 1).
Arm/Group | Placebo: Participated in Graduate OLE | Placebo: No Participation in Graduate OLE | Gantenerumab: Participated in Graduate OLE | Gantenerumab: No Participation in Graduate OLE
All-Cause Mortality (participants affected / at risk) | 0/14 | 5/691 | 2/29 | 4/647
Serious Adverse Events (participants affected / at risk) | 2/14 | 72/691 | 4/29 | 54/647
Other Adverse Events (participants affected / at risk) | 13/14 | 395/691 | 21/29 | 358/647
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo: Participated in Graduate OLE (N=14) | Placebo: No Participation in Graduate OLE (N=691) | Gantenerumab: Participated in Graduate OLE (N=29) | Gantenerumab: No Participation in Graduate OLE (N=647)
Anaemia (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 2 (2)
Atrial fibrillation (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Atrioventricular block complete (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cardiac arrest (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cardio-respiratory arrest (Cardiac disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cor pulmonale acute (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tachycardia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Meniere's disease (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal fistula (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Anal ulcer (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chest pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Generalised oedema (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pain (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pyrexia (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cholecystitis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 0 (0) | 3 (3) | 0 (0) | 3 (3)
COVID-19 pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Diverticulitis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Escherichia urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Pneumonia (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 1 (1)
Pneumonia aspiration (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 2 (2)
Skin infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 2 (2) | 0 (0) | 1 (1)
Wound infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Concussion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 4 (4) | 1 (1) | 4 (4)
Femur fracture (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Fracture displacement (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Head injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hip fracture (Injury, poisoning and procedural complications) | 0 (0) | 3 (4) | 0 (0) | 1 (1)
Humerus fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Radius fracture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Road traffic accident (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Subdural haemorrhage (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Toxicity to various agents (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper limb fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Wound (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Troponin increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malnutrition (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Chronic myeloid leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastric leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Glioblastoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatobiliary neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Invasive breast carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Melanoma recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Dysstasia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Epileptic encephalopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Hydrocephalus (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
Motor dysfunction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Seizure (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural hygroma (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Thalamus haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 2 (2)
Upper motor neurone lesion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Vasogenic cerebral oedema (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Agitation (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Confusional state (Psychiatric disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Delirium (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Calculus bladder (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ovarian cyst (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Vaginal prolapse (Reproductive system and breast disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 5 (5) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Aortic dissection (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Deep vein thrombosis (Vascular disorders) | 0 (0) | 3 (3) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Orthostatic hypotension (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral arterial occlusive disease (Vascular disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peripheral artery aneurysm (Vascular disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo: Participated in Graduate OLE (N=14) | Placebo: No Participation in Graduate OLE (N=691) | Gantenerumab: Participated in Graduate OLE (N=29) | Gantenerumab: No Participation in Graduate OLE (N=647)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1) | 4 (4) | 0 (0) | 2 (2)
Arrhythmia (Cardiac disorders) | 1 (1) | 0 (0) | 2 (3) | 0 (0)
Cardiac failure chronic (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Hydrocele (Congenital, familial and genetic disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dry eye (Eye disorders) | 1 (1) | 3 (3) | 0 (0) | 2 (2)
Anal incontinence (Gastrointestinal disorders) | 1 (1) | 5 (5) | 0 (0) | 6 (7)
Colitis (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 14 (14) | 0 (0) | 13 (13)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 13 (15) | 0 (0) | 17 (20)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 2 (2) | 1 (1) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 1 (1) | 10 (15) | 0 (0) | 23 (29)
Fatigue (General disorders) | 0 (0) | 17 (20) | 2 (2) | 10 (10)
Injection site reaction (General disorders) | 3 (5) | 63 (157) | 1 (10) | 80 (266)
Bacteriuria (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
COVID-19 (Infections and infestations) | 3 (3) | 114 (116) | 3 (3) | 90 (92)
Dacryocystitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Dermatophytosis of nail (Infections and infestations) | 1 (1) | 3 (3) | 0 (0) | 0 (0)
Gastroenteritis (Infections and infestations) | 1 (1) | 4 (4) | 0 (0) | 6 (7)
Nasopharyngitis (Infections and infestations) | 1 (2) | 25 (28) | 0 (0) | 29 (30)
Pelvic inflammatory disease (Infections and infestations) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Pharyngitis (Infections and infestations) | 1 (1) | 4 (4) | 1 (1) | 1 (1)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 1 (1) | 2 (2) | 1 (1)
Sinusitis (Infections and infestations) | 1 (1) | 4 (5) | 0 (0) | 0 (0)
Urinary tract infection (Infections and infestations) | 3 (9) | 30 (38) | 1 (2) | 37 (52)
Urosepsis (Infections and infestations) | 1 (3) | 0 (0) | 0 (0) | 0 (0)
Contusion (Injury, poisoning and procedural complications) | 3 (4) | 20 (21) | 2 (2) | 13 (35)
Fall (Injury, poisoning and procedural complications) | 4 (7) | 50 (67) | 6 (10) | 59 (92)
Head injury (Injury, poisoning and procedural complications) | 1 (1) | 5 (5) | 1 (1) | 4 (4)
Procedural pain (Injury, poisoning and procedural complications) | 2 (2) | 2 (4) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 2 (2) | 2 (3)
Wrist fracture (Injury, poisoning and procedural complications) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Vitamin B12 decreased (Investigations) | 0 (0) | 11 (12) | 2 (2) | 5 (5)
Vitamin B12 deficiency (Metabolism and nutrition disorders) | 0 (0) | 14 (14) | 2 (2) | 15 (15)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 25 (26) | 1 (1) | 33 (39)
Arthritis (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 15 (16) | 2 (2) | 32 (36)
Myalgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 3 (3) | 2 (2) | 3 (3)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1) | 6 (6) | 1 (1) | 5 (6)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
Amyloid related imaging abnormality-microhaemorrhages and haemosiderin deposits (Nervous system disorders) | 1 (1) | 21 (22) | 0 (0) | 7 (7)
Amyloid related imaging abnormality-oedema/effusion (Nervous system disorders) | 5 (5) | 67 (76) | 3 (4) | 16 (17)
Cerebral haemorrhage (Nervous system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 23 (27) | 4 (5) | 22 (23)
Dysarthria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 1 (1) | 33 (41) | 1 (1) | 24 (46)
Ischaemic stroke (Nervous system disorders) | 1 (2) | 3 (3) | 0 (0) | 1 (1)
Migraine (Nervous system disorders) | 1 (1) | 3 (3) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Somnolence (Nervous system disorders) | 1 (1) | 8 (10) | 2 (2) | 3 (3)
Aggression (Psychiatric disorders) | 1 (2) | 8 (8) | 1 (1) | 3 (3)
Anxiety (Psychiatric disorders) | 1 (1) | 11 (11) | 1 (1) | 14 (14)
Confusional state (Psychiatric disorders) | 1 (1) | 11 (12) | 0 (0) | 9 (13)
Delusion (Psychiatric disorders) | 0 (0) | 2 (2) | 2 (2) | 4 (4)
Depression (Psychiatric disorders) | 0 (0) | 12 (12) | 2 (2) | 5 (5)
Hallucination (Psychiatric disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Insomnia (Psychiatric disorders) | 1 (1) | 16 (17) | 1 (1) | 16 (16)
Irritability (Psychiatric disorders) | 0 (0) | 5 (5) | 2 (2) | 4 (4)
Bladder irritation (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Stress urinary incontinence (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Urinary incontinence (Renal and urinary disorders) | 1 (1) | 6 (6) | 0 (0) | 4 (4)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 3 (3) | 1 (1) | 1 (2)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
Dermatosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 4 (4) | 0 (0) | 8 (8)
Rash (Skin and subcutaneous tissue disorders) | 1 (1) | 11 (12) | 2 (2) | 9 (12)
Arteriosclerosis (Vascular disorders) | 1 (1) | 4 (4) | 0 (0) | 1 (1)
Hypertension (Vascular disorders) | 3 (3) | 14 (15) | 2 (2) | 19 (22)
Hypertensive crisis (Vascular disorders) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Hypotension (Vascular disorders) | 2 (2) | 10 (10) | 0 (0) | 11 (11)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Study being conducted under this Agreement is part of the Overall Study. Investigator is free to publish in reputable journals or to present at professional conferences the results of the Study, but only after the first publication or presentation that involves the Overall Study. The Sponsor may request that Confidential Information be deleted and/or the publication be postponed in order to protect the Sponsor's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-05-11): https://cdn.clinicaltrials.gov/large-docs/53/NCT04374253/Prot_000.pdf
  • Statistical Analysis Plan (2023-11-30): https://cdn.clinicaltrials.gov/large-docs/53/NCT04374253/SAP_001.pdf